CLINICAL TRIAL: NCT01382940
Title: A Multicenter, Open-label, Single-arm Study to Evaluate the Safety Administering Rituximab at a More Rapid Infusion Rate in Patients With Rheumatoid Arthritis
Brief Title: A Study on The Safety of Administering Rituximab at A More Rapid Rate in Patients With Rheumatoid Arthritis
Acronym: RATE-RA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25641
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Results first posted 2014-02-19 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate; Methylprednisolone; Acetaminophen; Histamine Antagonists

ARMS (1):
- Rituximab (Experimental): Rituximab intravenous (IV) infusions were administered over a 4.25-hour period on Day 1, and over a 2-hour period on Day 15 (first course) and on Days 168 and 182 (second course). All participants continued to receive methotrexate as prescribed by their treating physician. Premedication included methylprednisolone, an antihistamine and acetaminophen.
  Interventions: Drug: rituximab; Drug: methotrexate; Drug: methylprednisolone; Drug: acetaminophen; Drug: antihistamine

INTERVENTIONS:
Drug: rituximab — 1000 mg in 250 mL intravenous infusion
  Other Names: Rituxan®; MabThera®
Drug: methotrexate — 10 to 25 mg/week (oral or parenteral)
Drug: methylprednisolone — 100 mg methylprednisolone administered by slow intravenous infusion at least 30 minutes prior to the start of each study drug infusion
Drug: acetaminophen — 1 gram acetaminophen administered orally 30 to 60 minutes prior to the start of each study drug infusion
Drug: antihistamine — 50 mg diphenhydramine hydrochloride or equivalent dose of alternate antihistamine administered orally 30 to 60 minutes prior to the start of each study drug infusion

SUMMARY:
This study was designed to evaluate the safety of administering rituximab at a more rapid infusion rate in patients with moderate to severe rheumatoid arthritis who have had an inadequate response to biopharmaceuticals that treat diseases by interfering with tumor necrosis factor (anti-TNF therapies), and were receiving methotrexate therapy for more than eight weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult patients, ≥ 18 years of age
* Rheumatoid arthritis of ≥ 6 months duration, diagnosed according to the revised 1987 American College of Rheumatology criteria
* Inadequate response to at least one approved anti-TNF agent (adalimumab, etanercept, infliximab, golimumab, or certolizumab)
* Patients who have received 1 to 2 prior courses of rituximab (RTX) may be enrolled, provided their most recent course of RTX occurred over 6 months but no more than 9 months prior to baseline. The RTX dosage must have been two 1000 mg infusions per course administered at the standard approved rate
* Methotrexate treatment between 10 and 25 mg/week (oral or parenteral) for at least 8 weeks immediately prior to baseline

Key Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned surgery within 6 months following baseline
* Rheumatic autoimmune disease other than rheumatoid arthritis
* Functional class IV as defined by American College of Rheumatology (ACR) criteria
* Prior history of or current inflammatory joint disease other than rheumatoid arthritis
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies
* Previous serious infusion reaction to any prior biologic therapy
* Known active current or history of recurrent infection
* Evidence of chronic hepatitis B or C infection
* Pregnant or lactating women
* Body weight of > 150 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2011-07-26 (Actual); Primary Completion 2013-01-06 (Actual); Study Completion 2013-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (86):
- United States (86):
  - Uni Of Alabama,Birmingham; Medicine - Rheumatology, Birmingham, Alabama
  - Clnical & Translational Reseach Center for Alabama, PC, Tuscaloosa, Alabama
  - ArthroCare, Arthritis Care; and Research P.C., Gilbert, Arizona
  - Valley Arthritis Care, Phoenix, Arizona
  - Catalina Pointe Rheumatology, Tucson, Arizona
  - Medvin Clinical Research, Covina, California
  - Triwest Research Associates, La Mesa, California
  - Medvin Clinical Research, Los Angeles, California
  - Brigid Freyne-Private Practice; Internal Medicine, Rheum, Murrieta, California
  - Desert Medical Advances; Rheumatology, Palm Desert, California
  - San Diego Arthritis Med Clnc, San Diego, California
  - Pacific Arthritis Ctr Med Grp, Santa Maria, California
  - Inland Rheumatology; Clinical Trials, Inc., Upland, California
  - Medvin Clinical Research, Whittier, California
  - Arthritis Assoc & Osteoporosis; Ctr of Colorado Springs, Colorado Springs, Colorado
  - Denver Arthritis Clinic, Denver, Colorado
  - Rheum & Internal Med Assoc-Bri, Bridgeport, Connecticut
  - Arthritis & Osteoporosis Center Pc, Hamden, Connecticut
  - Rheumatolgy Consultants of Deleware, Lewes, Delaware
  - Javed Rheumatology Associates, Inc., Newark, Delaware
  - Arthritis & Rheumatism; Disease Specialities, Aventura, Florida
  - Florida Arthritis Center, PI, Lake Mary, Florida
  - Omega ResearchConsultants LLC, Orlando, Florida
  - Millenium Research, Ormond Beach, Florida
  - Arthritis Center Palm Harbor, Palm Harbor, Florida
  - Arthritis Rsrch of Florida, Inc., Palm Harbor, Florida
  - Center For Arthritis; Research Dept, South Miami, Florida
  - University of South Florida, Tampa, Florida
  - Florida Medical Clinic; Clinical Research, Zephyrhills, Florida
  - Parris & Associates, Lawrenceville, Georgia
  - St. Luke's Intermountain Research Center, Boise, Idaho
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Quad City Rheumatology, Sc, Moline, Illinois
  - Physician'S Clinic of Iowa, Cedar Rapids, Iowa
  - Bluegrass Comm Research, Inc., Lexington, Kentucky
  - Klein & Associates, M.D. P.A., Cumberland, Maryland
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - St. Luke's Hospital Association of Duluth, Duluth, Minnesota
  - Arthritis and Osteoporosis; Treatment and Research Center, Flowood, Mississippi
  - Jackson Arthritis Clinic, Flowood, Mississippi
  - North Mississippi Med Clinics, Inc., Tupelo, Mississippi
  - David S Rosenberg, Florissant, Missouri
  - Arthritis Center of Reno, Reno, Nevada
  - Rheumatology Research Group, Lebanon, New Hampshire
  - Rheumatology Associates Of New Jersey, Teaneck, New Jersey
  - The Center for Rheumatology, Albany, New York
  - Arthritis & Osteoporosis Center, Brooklyn, New York
  - NYU Center for Musculoskeletal Care, New York, New York
  - Buffalo Rheumatology Associates, Orchard Park, New York
  - Office of Premier Chatpar Md, Plainview, New York
  - Aair Research Center, Rochester, New York
  - Rheumatology Associates of Long Island, Smithtown, New York
  - Arthritis Health Associates; Clinical Research, Syracuse, New York
  - Arth&OsteoConsof theCarolinas-Charlotte, Charlotte, North Carolina
  - Box Arthritis & Rheumatology, Charlotte, North Carolina
  - Carolina Bone & Joint P.A., Charlotte, North Carolina
  - Physicians East Pa, Greenville, North Carolina
  - Shanahan Rheumatology & Immunology, PLLC, Raleigh, North Carolina
  - Crystal Arthritis Center, Inc., Akron, Ohio
  - CarePoint East, Columbus, Ohio
  - Stat Research, Inc, Dayton, Ohio
  - Paramount Medical Research, Middleburg Heights, Ohio
  - LION Research, Norman, Oklahoma
  - Arthritis and Rheumatology; Center of Oklahoma PLLC, Oklahoma City, Oklahoma
  - East Penn Rheumatology Associates, Pc, Bethlehem, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Pivotal Clinical Research, Llc, Perkasie, Pennsylvania
  - Arthritis Group, Philadelphia, Pennsylvania
  - Rheumatic Disease Associates; Clinical Research Unit, Willow Grove, Pennsylvania
  - Clinical Research Center of Reading, Wyomissing, Pennsylvania
  - Pennsylvania Regional Center for Arthritis and Osteoporosis Research, Wyomissing, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - Rheumatology Associates, Charleston, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Ramesh Gupta - PP, Memphis, Tennessee
  - Amarillo Center For Clinical Research, Amarillo, Texas
  - Lovelace Scientific Resources Inc., Austin, Texas
  - Adriana Pop-Moody MD Clinic PA, Corpus Christi, Texas
  - Arthritis Centers of Texas, Dallas, Texas
  - Southwest Rheumatology, Mesquite, Texas
  - Arthritis Clinic of Northern Virginia, Arlington, Virginia
  - Apex Clinical Research, Kennewick, Washington
  - Seattle Arthritis Clinic, Seattle, Washington
  - Arthritis Northwest, Spokane, Spokane, Washington
  - Cedar Medical Center, Tacoma, Washington
  - Rheumatic Disease Center, Glendale, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab
Started | 351
Received Day 1 Infusion | 351
Received Day 15 Infusions | 341
Received Day 168 Infusion | 290
Received Day 182 Infusion | 278
Completed | 278
Not Completed | 73
Not completed — Adverse Event | 19
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 7
Not completed — Withdrawal by Subject | 23
Not completed — Protocol Violation | 20

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 351
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 279
  Male | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Any Infusion-related Reaction (IRR) Associated With the Second Rituximab Infusion
Description: The primary criterion for assessing safety of the faster infusion was the incidence of infusion related reaction (IRRs). IRRs were adverse events (AEs) that occurred within 24 hours of beginning infusion that were among a pre-specified list of preferred terms from the Medical Dictionary for Regulatory Activities (MedDRA). "Incidence" is defined as the percentage of participants experiencing an IRR.
Time Frame: Within 24 hours of beginning infusion on Day 15
Population: All randomized participants who received infusion at the faster rate on Day 15. Four participants who received the Day 15 rituximab infusion were excluded from the primary analysis population because their infusion rates could not be determined.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 337
percentage of participants | 6.5 (6.5) [4.1 to 9.7]

2. Secondary Outcome: Percentage of Participants Experiencing Any Serious IRR (SIRR) Associated With the Second Rituximab Infusion
Description: A serious infusion-related reaction (SIRR) is an IRR that meets the definition of a serious adverse event. A serious adverse event (SAE) is any experience that suggests a significant hazard, contraindication, side effect or precaution.
Time Frame: Within 24 hours of beginning infusion on Day 15
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 337
percentage of participants | 0.0 [0.0 to 1.1]

3. Secondary Outcome: Percentage of Participants Experiencing Any IRR or SIRR Associated With the Third Rituximab Infusion
Description: IRRs are AEs that occurred within 24 hours of beginning infusion that were included on a pre-specified list of MedDRA preferred terms, and an SIRR is an IRR that suggests a significant hazard, contraindication, side effect or precaution.
Time Frame: Within 24 hours of beginning infusion on Day 168
Population: All randomized participants who received infusion at the faster rate on Day 168. One participant received the Day 168 rituximab infusion at the labeled rate rather than at the faster rate and was excluded from the analysis population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 289
percentage of participants
  Any IRR | 5.9 [3.5 to 9.3]
  Any SIRR | 0.0 [0.0 to 1.3]

4. Secondary Outcome: Percentage of Participants Experiencing Any Common Toxicity Criteria (CTC) Grade 3 or 4 Adverse Events (AEs) Associated With the Second Rituximab Infusion
Description: The intensity of AEs were graded on a 5-point scale (Grade 1 to 5) according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v. 4.0), where Grade 1 indicates "Mild" severity and Grade 5 indicates "Death". The CTCAE defines Grades 3 and 4 as follows: - Grade 3 means "Severe", indicating considerable interference with the patient's daily activities; medical intervention/therapy required; and hospitalization possible. - Grade 4 means "Life-threatening, Disabling", based on extreme limitation in activity; significant medical intervention/therapy required, and hospitalization probable.
Time Frame: Within 24 hours of beginning infusion on Day 15
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 337
percentage of participants | 0.6 [0.1 to 2.1]

5. Secondary Outcome: Percentage of Participants Experiencing the Stopping, Slowing or Interrupting of the Second Rituximab Infusion
Description: Participants who experienced a moderate or serious IRR had their infusion interrupted immediately and received aggressive symptomatic treatment. The CTCAE includes the following severity descriptions: - "Moderate" means mild to moderate interference with the patient's daily activities, no or minimal medical intervention/therapy required; - "Severe" means considerable interference with the patient's daily activities, medical intervention/therapy required, hospitalization possible. If the IRR was moderate, the infusion was not to be restarted before all the symptoms disappeared, and then at half the rate. If the participant tolerated the reduced rate for 30 minutes, the infusion rate was increased to the next rate on the protocol-specified infusion schedule. If the symptoms did not resolve with treatment, the participant was withdrawn from the treatment period of the study. Participants who experienced a severe IRR to rituximab treatment were discontinued from the study.
Time Frame: During the infusion (a 2-hour period) on Day 15
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 337
percentage of participants | 3.9 [2.1 to 6.5]

6. Secondary Outcome: Percentage of Participants Experiencing Any Common Toxicity Criteria (CTC) Grade 3 or 4 Adverse Events (AEs) Associated With the Third Rituximab Infusion
Description: The intensity of AEs experienced within 24 hours of beginning infusion were graded on NCI's CTCAE (v. 4.0) intensity scale from Grade 1 ("Mild") to Grade 5 ("Death"). Grade 3 AEs are "Severe" and Grade 4 AEs are "Life-threatening, Disabling".
Time Frame: Within 24 hours of beginning infusion on Day 168
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 289
percentage of participants | 0.0 [0.0 to 1.3]

7. Secondary Outcome: Percentage of Participants Experiencing the Stopping, Slowing or Interrupting of the Third Rituximab Infusion
Description: as for outcome 5
Time Frame: During the infusion (a 2-hour period) on Day 168
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 289
percentage of participants | 6.6 [4.0 to 10.1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at each visit and during a follow-up telephone visit four weeks after the last rituximab infusion (Day 210).
Description: The safety evaluable population included all participants who received rituximab during the study and had at least one safety assessment during or after the rituximab infusion.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 30/351
Other Adverse Events (participants affected / at risk) | 37/351
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=351)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Device breakage (General disorders) | 1
Chest discomfort (General disorders) | 1
Pneumonia (Infections and infestations) | 4
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Complex partial seizures (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=351)
Upper Respiratory Tract Infection (Infections and infestations) | 19
Headache (Nervous system disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.